CLINICAL TRIAL: NCT04020952
Title: Effect of Archwire Gauge on the Rate of Canine Retraction in Adults: A Randomized Clinical Trial
Brief Title: Effect of Archwire Gauge on the Rate of Canine Retraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aml Saeed Mohamed Abdel qader, masters degree student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 334
Record Dates: First submitted 2019-07-09; First posted 2019-07-16 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Canine Retraction
Keywords: canine retraction; archwire gauge

STUDY DESIGN:
Intervention Model Description: Three groups of patients each receives different wire gauge during canine retraction phase during space closure.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor is not informed about the gauge of the wire used for patients
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- st.st 0.019×0.025" wire (Active Comparator)
  Interventions: Other: st.st 0.019×0.025" wire
- st.st 0.016×0.022" wire (Experimental)
  Interventions: Other: st.st 0.016×0.022" wire
- st.st 0.017×0.025" wire (Experimental)
  Interventions: Other: st.st 0.017×0.025" wire

INTERVENTIONS:
Other: st.st 0.019×0.025" wire — rectangular stainless steel wire that will be used during canine retraction after first premolars extraction
  Arms: st.st 0.019×0.025" wire
Other: st.st 0.016×0.022" wire — rectangular stainless steel wire that will be used during canine retraction after first premolars extraction
  Arms: st.st 0.016×0.022" wire
Other: st.st 0.017×0.025" wire — rectangular stainless steel wire that will be used during canine retraction after first premolars extraction
  Arms: st.st 0.017×0.025" wire

SUMMARY:
trial will be done to evaluate the effect of archwire gauge on the rate of canine retraction, canine tip and torque, root resorption and loss of anchorage in maxillary dental protrusion cases requiring first premolars extraction.

DETAILED DESCRIPTION:
Three working archwires of different gauges will be used during canine retraction; st.st 0.019×0.025" as a comparator, st.st 0.016×0.022" and st.st 0.017×0.025" wires as interventions. after levelling and alignment till reaching the working archwire, it will be left in place for a month then maxillary first premolars will be extracted and base line records will be taken(digital models, digital periapical radiographs and panorama). digital models will be taken monthly to measure rate of canine retraction for 6 months. after 6 month evaluation of anchorage loss, change in canine tip and torque will be done on last obtained digital model , panorama will be taken to evaluate the change in canine tip and digital periapical radiograph will be taken and compared with the preretraction radiograph to evaluate amount of root resorption.

ELIGIBILITY:
Inclusion Criteria:

* Adult females (age range 18-28 years old).
* Maxillary dental protrusion indicating first premolars extraction.
* Full permanent dentition (not necessitating third molars).

Exclusion Criteria:

* Patients having systemic diseases or on medications that would affect tooth movement.
* Active periodontal disease or obvious bone resorption in maxillary arch.
* Patients with habits that are detrimental to dental occlusion (thumb sucking, tongue thrusting … etc.).
* Previous orthodontic treatment.
* Missing teeth.

Ages: 16 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — adult female patients
Enrollment: 18 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
rate of canine retraction | 6 months
  the distance that canine moved every month

SECONDARY OUTCOMES:
change in canine tip | 6 months
  change in canine crown tipping to certain reference plane with the aid of cone beam computed tomography
change in canine torque | 6 months
  change in canine crown and root torque to certain reference plane with the aid of cone beam computed tomography
loss of molar anchorage | 6 months
  assess from digital models if there is change in mesio-distal position of maxillary first molar
amount of canine root resorption | 6 months
  assess amount of root resorption (if occurred) with the aid of cone beam computed tomography

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry, Cairo University, Cairo, Egypt

REFERENCES:
- [Derived] Abdelkader ASM, Abd El-Ghafour M, Dehis HM, El Sharaby FA, Labib AH. Effect of archwire size on the rate of canine retraction in adult women : A randomized clinical trial. J Orofac Orthop. 2025 Mar 25. doi: 10.1007/s00056-025-00577-y. Online ahead of print. PMID 40131446